CLINICAL TRIAL: NCT02862925
Title: Introducing Fetal Scalp Stimulation as an Adjunct to Intermittent Auscultation in Low-Resource Settings.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Fulbright (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00070952; R25TW009337 (NIH)
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-04

CONDITIONS: Fetal Distress; Stillbirth; Birth Asphyxia; Acidosis
Keywords: fetal monitoring; cesarean delivery; obstetrics; midwifery; developing countries
MeSH Terms: conditions — Fetal Distress; Stillbirth; Asphyxia Neonatorum; Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-Intervention (No Intervention): A consecutive sample of 350 patients will be collected. After informed consent, data will be abstracted from the patient's record including day and time of delivery, method of delivery, parity, gestational age, meconium presence, heart rate abnormality and induction methods. For CD, the following data will be collected: decision-to-delivery time, Partogram adherence, time of each FSST, Apgar score, date and time of delivery and Comorbidities such as: Hypertension-spectrum disorders, Malaria, Postpartum Hemorrhage, Macrosomia, History of CD, Diabetes, Sickle Cell, and HIV status.
- Post-intervention (Experimental): The study will take place on the labor ward at KCMC in Moshi, Tanzania. It will involve women who present to the labor ward in labor or who undergo an induction of labor. A consecutive sample of 350 patients will be collected. Study investigators will be present for 24 hours a day, 7 days a week on a rotating schedule during the enrollment period. All patients who fit inclusion and exclusion criteria will be approached if they are deemed medically stable.
  Interventions: Procedure: Fetal Scalp Stimulation

INTERVENTIONS:
Procedure: Fetal Scalp Stimulation — During a routine vaginal exam, if there is concern for fetal distress based on local definitions, the midwife will gently stroke the fetal head with her finger. She will then observe for a rise in the fetal heart rate as observed by the Doppler monitor. A rise to above 15 beats per minute above the baseline is termed an "acceleration" and NEGATIVE test. Absence of an acceleration is a POSITIVE test and reason for intervention.
  Arms: Post-intervention

SUMMARY:
This study is a pilot study taking place in Moshi, Tanzania at the Kilimanjaro Christian Medical Centre (KCMC). The study aims to introduce fetal scalp stimulation into the intermittent auscultation protocols at KCMC, and to validate whether or not a handheld Doppler device can perform the fetal scalp stimulation test accurately.

DETAILED DESCRIPTION:
Background:

Each year an estimated 2.6 million stillbirths occur globally. Nearly half, 1.2 million, of these occur intrapartum and an additional 650,000 children are born alive but die soon after birth due to birth asphyxia which is caused by hypoxia during labor. The vast majority of these deaths occur in low- and middle-income countries (LMICs). In high-income countries, obstetric providers utilize electronic fetal monitoring (EFM) to monitor fetuses during labor, but controversy surrounds implementing this technology in LMICs. What observing EFM patterns has taught us is that fetuses that respond to scalp stimulation with a rise in their heart rate are essentially guaranteed to be well oxygenated. This physiologic phenomenon, known as the fetal scalp stimulation test (FSST), has potential to improve fetal monitoring in LMICs, but it has never been studied using Doppler technology. This study aims to collect information about the prevalence of fetal distress in an obstetric referral hospital, to test the sensitivity and specificity of FSST with a Doppler device, and to collect pilot data using FSST as an adjunct to improve fetal monitoring. The outcome of the study would be to identify a trend in cesarean delivery rate reduction, intrapartum stillbirth, and birth asphyxia.

The vast majority of acute intrapartum-related morbidity and mortality occurs in low- and middle-income countries (LMIC) where the care of mothers and fetuses during labor remains under studied as is our understanding of how to implement and evaluate programs that address the delivery of quality care. Providing safe and effective obstetric care requires the development of processes that are appropriate for each clinical setting considering resources, burden of disease, and cultural factors as well as implementing those processes in an effective way so that they become standard practice over time. Internationally midwives employ intermittent auscultation (IA) to monitor fetuses with Pinard stethoscopes or Doppler devices. In high-resource settings providers rely on computerized electronic fetal monitoring (EFM) to identify signs of fetal acidosis, although this has not been shown superior to IA. Recently, the Federation International of Gynecology and Obstetrics published recommendations for adjunctive tests to fetal monitoring, but the recommendations were limited to the high-resource EFM paradigm. On this subject, an expert on fetal physiology from Nigeria stated, "it is imperative that appropriate diagnostic and management modalities for fetal hypoxia be available and accessible. This is the only way the burden of perinatal morbidity and mortality can be reduced." Currently, fetal scalp stimulation (FSST) is the only low-cost, validated, adjunctive test that could be used to this end in the majority world, but it has not been studied for this purpose.

STATEMENT OF THE PROBLEM Tanzania ranks as the 9th worst country for stillbirth globally experiencing 47,100 losses in 2015. Fetal monitoring at Kilimanjaro Christian Medical Center (KCMC) in Moshi, Tanzania, and countless labor wards around the world, is limited by the inability to accurately identify fetal acidosis in laboring patients. Misdiagnosis leads either to excess cesarean delivery (CD) or excess asphyxiated births. The study hypothesis is that implementing fetal scalp stimulation test (FSST) into labor protocols will reduce CD rates and improve neonatal outcomes leading to a reduction in maternal and neonatal mortality. Proving this will require a large randomized-controlled trial (RCT). The necessary first step is a proof-of-concept, feasibility study that will provide pilot data and inform future efforts.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age ≥ 37 weeks
* Singleton gestation
* Cephalic presentation
* First stage of labor
* Fetal distress diagnosed in the labor ward by either FHR >160 or <110, and/or grade 2-3 meconium-stained liquor

Exclusion Criteria:

* Chorioamnionitis
* Known fetal anomaly
* Antepartum hemorrhage
* Eclampsia
* Other maternal/fetal factors precluding vaginal delivery

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 550 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by completion of all 3 study objectives | Day 1
Predicted fetal acidosis from cord blood pH (at thresholds of cord blood pH<7.0, 7.1, and 7.2) | Day 1
  The primary outcome is the sensitivity and specificity of the Doppler device to predict fetal acidosis based on the fetal scalp stimulation test.

SECONDARY OUTCOMES:
Fetal distress rate | Day 1
  The investigators plan to define the fetal distress rate at a large referral center in Tanzania
Change in cesarean delivery rate | baseline, post introduction of fetal scalp stimulation (during labour)
  The investigators plan to compare cesarean delivery rates before and after the introduction of fetal scalp stimulation to fetal monitoring protocols.

OTHER OUTCOMES:
Birth asphyxia/stillbirth rate | Day 1
NICU Admission Rate | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: John Schmitt, MD, Principal Investigator — Duke UMC, Duke Global Health Institute
Locations (1):
- Kilimanjaro Christian Medical Center, Moshi, Kilimanjaro, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visser GH, Ayres-de-Campos D; FIGO Intrapartum Fetal Monitoring Expert Consensus Panel. FIGO consensus guidelines on intrapartum fetal monitoring: Adjunctive technologies. Int J Gynaecol Obstet. 2015 Oct;131(1):25-9. doi: 10.1016/j.ijgo.2015.06.021. No abstract available. PMID 26433402
- [Background] Omo-Aghoja L. Maternal and fetal Acid-base chemistry: a major determinant of perinatal outcome. Ann Med Health Sci Res. 2014 Jan;4(1):8-17. doi: 10.4103/2141-9248.126602. PMID 24669324
- [Background] Clark SL, Gimovsky ML, Miller FC. The scalp stimulation test: a clinical alternative to fetal scalp blood sampling. Am J Obstet Gynecol. 1984 Feb 1;148(3):274-7. doi: 10.1016/s0002-9378(84)80067-8. PMID 6695974
- [Background] Clark SL, Gimovsky ML, Miller FC. Fetal heart rate response to scalp blood sampling. Am J Obstet Gynecol. 1982 Nov 15;144(6):706-8. doi: 10.1016/0002-9378(82)90441-0. PMID 7137256
- [Background] Skupski DW, Rosenberg CR, Eglinton GS. Intrapartum fetal stimulation tests: a meta-analysis. Obstet Gynecol. 2002 Jan;99(1):129-34. doi: 10.1016/s0029-7844(01)01645-3. PMID 11777523
- [Background] Rathore AM, Ramji S, Devi CB, Saini S, Manaktala U, Batra S. Fetal scalp stimulation test: an adjunct to intermittent auscultation in non-reassuring fetal status during labor. J Obstet Gynaecol Res. 2011 Jul;37(7):819-24. doi: 10.1111/j.1447-0756.2010.01442.x. Epub 2011 Mar 16. PMID 21410829
- [Derived] Goodman DM, Mlay P, Thielman N, Small MJ, Schmitt JW. Using fetal scalp stimulation with Doppler ultrasonography to enhance intermittent auscultation in low-resource settings: a diagnostic trial from Tanzania. BMC Pregnancy Childbirth. 2019 Feb 13;19(1):71. doi: 10.1186/s12884-019-2212-z. PMID 30760224
- See also: Sustainable Development Goals & Topics .:. Sustainable Development Knowledge Platform — https://sustainabledevelopment.un.org/topics